CLINICAL TRIAL: NCT03547882
Title: APEX- Addiction Treatment in Primary Care Expansion (PII 18-181)
Brief Title: Addiction Treatment in Primary Care Expansion
Acronym: APEX
Status: Withdrawn | Type: Observational
Why Stopped: Project ended in 2022 and evolved into another grant (VA PII 19-321 (050 HX003009))
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Eastern Colorado Health Care System (U.S. Federal Agency); University of Colorado, Denver (Other); University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: PIX 18-002; PII 18-181 (Other Grant/Funding Number: Quality Enhancement Research Initiative (QUERI))
Record Dates: First submitted 2018-04-24; First posted 2018-06-06 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Opioid Use Disorder (OUD); Chronic Pain
Keywords: Opioid; Buprenorphine; Naltrexone; methadone
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: None Retained — No Bio specimen collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Other: Target interviewees will be primary care providers at six facilities and their staff (e.g., nurse care managers).
- Patients: Ten interviews were conducted with VA patients receiving ORT.

SUMMARY:
The Veterans Health Administration (VA) is a national leader in addressing the twin epidemics of chronic pain and opioid use, misuse, and opioid use disorder (OUD); but important challenges remain. Both chronic pain and OUD are more common among Veterans compared to the general population.1 As the VA transitions toward a greater emphasis on non-opioid chronic pain treatments, improving access to OUD treatment will be critical for those Veterans with new diagnoses of OUD in the context of long-term opioid therapy. Strong evidence supports the treatment of OUD with medications, including naltrexone, buprenorphine, and methadone.2 Buprenorphine and naltrexone can be prescribed in primary care settings; OUD treatment in primary care is associated with decreased opioid use, higher quality of care, and improved quality of life.3-5 In partnership with VISN19 leadership, this project will address the priority goal of improving access to medication-assisted therapy for OUD treatment. The objective of the VISN Partnered Implementation Initiative startup phase (PHASE 1) is to implement and evaluate the evidence-based, effective practice of medication treatment of opioid use disorder in primary care settings. A subsequent PHASE 2 will study the implementation of strategies from PHASE 1 across the entire VISN19. The investigators propose two specific aims:

Aim 1: Evaluate the implementation and impact of a multifaceted provider support initiative at two VA medical centers and four community-based clinics in VISN19 using the integrated-Promoting Action on Research Implementation in Health Services (i-PARIHS) implementation framework. The multifaceted initiative will leverage existing VA and VISN resources (including e-consults, telementoring and telehealth) to facilitate improved access to OUD treatment in primary care.

Aim 2: Create an interactive implementation toolkit with guidance on facilitation and incentive strategies and resources for broader dissemination across the VISN and VA.

DETAILED DESCRIPTION:
Among Veterans receiving healthcare from the Veterans Health Administration (VA), there has been sharp rise in the number of veterans diagnosed with opioid use disorder (OUD). In 2013, 25,031 Veterans had OUD and in 2017, Veterans with OUD nearly tripled to 69,142.6 As the largest direct provider of addiction treatment nationally, VA has taken steps to increase access to medication treatment for OUD, which is recognized as an essential component of evidence-based care.

The treatment of OUD involves several FDA-approved, VA formulary medications including naltrexone, methadone, and buprenorphine/naloxone and buprenorphine (hereafter collectively termed buprenorphine). Strong evidence supports the treatment of OUD with medications, and they are the "gold standard" treatments for OUD. Medications for OUD have been shown to substantially decrease risk for all-cause mortality and overdose mortality in people with opioid use disorder. Unlike methadone, buprenorphine for OUD can be prescribed in office-based settings such as primary care, and buprenorphine delivered in primary care is associated with decreased opioid use, higher quality of care, and improved quality of life. Medication treatment includes dispensation of methadone and buprenorphine in licensed opioid treatment programs (OTPs) and prescriptions of buprenorphine and naltrexone in office-based settings. Because there are only 32 licensed OTPs in the VA, buprenorphine and naltrexone prescriptions are the means to improve access to medication treatment for Veterans with OUD. Uptake of medication treatment, however, has been slow and uneven in the VA. In 2017, 35% of Veterans diagnosed with OUD had received OUD medications.

In VISN19, rates of OUD and OUD treatment are low and heterogeneous across facilities and compared with the national average (35%), fewer patients with OUD are on OUD medications (21%) in VISN19. Multiple initiatives have been instituted to improve access to medication treatment for Veterans with OUD, particularly in non-specialty office-based settings. In 2007, VA introduced the Buprenorphine in the VA Initiative (BIV; Director Gordon), a national consult service, which aimed to improve care processes and patient outcomes associated with buprenorphine. In 2010, VA unrolled Academic Detailing program in which pharmacy specialists take on high-priority pharmaceutical education campaigns. An Academic Detailing campaign specifically targeting the treatment of opioid use disorder was initiated in 2017. Further improving access to evidence-based medication treatment of OUD remains a priority for VA and VISN19.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include health care providers at 2 main VA facilities and four VA community based outpatient clinics
* VA patients receiving ORT

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: VA Medical Providers and VA patients receiving ORT
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who receive mediation assisted treatment for opioid use disorder (by facility and community based clinic) | 12 Months
  Electronic health record and Administrative data will be pulled to assess outcomes
Ratio of patients receiving medication assisted treatment for opioid use disorder to the number of patients with opioid use disorder (by facility and community based clinic) | 12 Months
  Electronic health record and Administrative data will be pulled to assess outcomes
Change in number of providers prescribing medication assisted treatment for opioid use disorder and patients receiving medication assisted treatment (by facility) | baseline through 1 year
  Interviews to stakeholders facilitated by field note review will be conducted to examine facilitators and barriers of implementation
Patients receiving medication assisted treatment (by facility) | 12 Months
  The investigators will be using the VA Academic Detailing Data Tool System which includes different measures with real time patient tracker to identify patients receiving medication assisted treatment.
  By using different dashboards the investigators will be pulling number of patients with buprenorphine treatment and the number of OUD patients with OUD pharmacotherapy from this dashboards.

CONTACTS AND LOCATIONS:
Overall Officials: Adam J. Gordon, MD MPH, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT; Joseph W Frank, MD MPH, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (2):
- United States (2):
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No